CLINICAL TRIAL: NCT05722613
Title: Diagnostic Potential of the Salivary (miRNAs - 146-a, 186, IL-1ß, and IL- 10) to Differentiate Statuses of Periodontitis: A Case-Control Study
Brief Title: Diagnostic Potential of the Salivary Biomarkers to Differentiate Statuses of Periodontitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Zainab Jalil Raheem, principal invstigator, University of Baghdad
Other Study IDs: 527622
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Periodontitis
Keywords: periodontitis; saliva; case control
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- (Group A) periodontally healthy as a control: BOP <10%, PPD ≤ 3mm, intact periodontium (no probing attachment loss).
- (Group B) periodontitis currently unstable: Generalized periodontitis, currently unstable (PPD ≥ 5mm or PPD at ≥ 4mm with BOP).
- (Group C)periodontitis currently stable .: Generalized periodontitis, currently stable (BOP < 10 % PPD ≤4 mm and no BOP at 4mm sites)

SUMMARY:
Periodontitis is a chronic inflammatory disease characterized by both dysbiosis of oral microbiota and proinflammatory events involving both cells and mediators from innate and adaptive immunity. These events lead to chronic inflammation of periodontal soft and hard tissues sharing many features with other chronic inflammatory diseases. These events lead to chronic inflammation of periodontal soft and hard tissues sharing many features with other chronic inflammatory diseases. Chronic inflammation is driven by various mediators, of which a significant part is attributed to the interactions within cytokine networks. While proinflammatory cytokines, including interleukin (IL) -1α, IL-1β, TNF-α, IL-6, and IL-17, contribute to acute and chronic inflammation and tissue injury, a second group with antagonist effects is formed by cytokines such as IL-10

DETAILED DESCRIPTION:
Diagnosis of Periodontitis represents the backbone of a successful periodontal treatment since the entire treatment plan, prognosis, and maintenance directly depend on the quality and precision of periodontal diagnosis. Since periodontal diagnostics is still based on clinical and radiological parameters providing limited therapeutic guidance, biomarkers have been introduced for the first time within the new classification of periodontal and peri-implant conditions as a first step towards the adoption of precision medicine concepts in periodontology. Saliva, as part of oral fluids, is an optimal biological fluid that contains locally and systemically derived mediators of periodontal disease (proteins, genetic/genomic biomarkers such as DNA and mRNA, and various metabolites that originate from the host and the bacteria) to serve as the diagnostic tool for periodontitis. The collection of saliva is safe, non-invasive, and simple, and saliva can be collected repeatedly with minimum discomfort to the patient. Single biomarker detection may not be effective enough for accurate diagnoses without false-positive or false-negative results. Periodontitis is a disease that involves complex interactions between bacteria and the host immune system. The combination of the host and bacteria-derived biomarkers, which reflect inflammation, soft tissue destruction, and bone destruction together, may be helpful in the diagnosis

ELIGIBILITY:
Inclusion Criteria:

1. Male and female systemically healthy patients.
2. Body mass index ≤ 30.
3. Have a minimum of 20 teeth with facial and lingual scorable surfaces.
4. Clinical criteria for periodontal health and periodontitis will be as follows :

1. Healthy periodontium (Group A): BOP <10%, PPD ≤ 3mm, intact periodontium (no probing attachment loss).

2. Periodontitis groups are defined as : i. Interdental CAL is detectable at ≥2 non-adjacent teeth, or ii. Buccal or oral CAL ≥3 mm with pocketing >3mm is detectable at ≥2teeth

Exclusion Criteria:

1. Patients who refused to participate in the study.
2. Individuals with dental implants.
3. Previous history of extensive periodontal therapy preceding 6 months or currently under active periodontal treatment.
4. Patients receiving antibiotic treatment or immunosuppressant medication within the last 3 months
5. Pregnant or lactating mothers.
6. Any symptoms of recent acute illness, e.g., COVID-19.
7. Tobacco use.
8. Active orthodontic therapy

   -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited from the Department of Periodontics, College of Dentistry, University of Baghdad.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
diagnosis | base line
  The primary outcomes will be determining salivary levels of (miRNAs 146-a, 186, IL-1β, and IL-10

CONTACTS AND LOCATIONS:
Overall Officials: zainab J Raheem, MSc, Principal Investigator — University of Baghdad
Locations (1):
- University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Raheem ZJ, Abdulbaqi HR. Diagnostic Potential of Salivary Interleukin-1beta and IL-10 for Distinguishing Periodontal Health From Periodontitis and Stable From Unstable Periodontitis: A Case-Control Study. Int J Dent. 2024 Oct 15;2024:8006278. doi: 10.1155/2024/8006278. eCollection 2024. PMID 39445112